CLINICAL TRIAL: NCT03017664
Title: An Improvement Project Towards Optimizing Nutrition Intervention With a Higher Protein and Calorie Pediatric Tube Feeding Formula
Brief Title: Improvement Project To Optimizing Nutrition With Higher Protein and Calorie Pediatric Tube Feeding
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 16.04.US.HCN
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Critically Ill Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RFG: Retrospective review of enteral feeding in pediatric ICU patients for up to 5 days
  Interventions: Other: Retrospective review of enteral tube feeding formula
- PFG: Pediatric ICU population to be fed a peptide-based enteral formula with higher protein and higher calories for up to 5 days
  Interventions: Other: Peptide-based enteral formula

INTERVENTIONS:
Other: Peptide-based enteral formula — Peptide-based, higher protein and higher calorie enteral formula
  Groups: PFG
Other: Retrospective review of enteral tube feeding formula — Enteral formula tube feeding will be retrospectively reviewed
  Groups: RFG

SUMMARY:
This quality improvement project will include a practice change based on national guidelines for the nutritional management of PICU patients.

DETAILED DESCRIPTION:
This quality improvement project will include a practice change based on national guidelines for the nutritional management of PICU patients. The primary aim of this quality improvement project is to better meet protein needs of ICU critically ill children

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-18 years old with enteral feeding access and anticipated to be fed for 5 days

Exclusion Criteria:

-

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-13 years with enteral feeding access
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Enteral formula volume | 5 days
  Daily total formula volume (mL) delivered

OTHER OUTCOMES:
Protein modular | 5 days
  yes/no; if yes, dose (g/mL) and schedule
Enteral feeding interruptions | 5 days
  yes/no; if yes, reason for interruption
Diarrhea | 5 days
  yes/no; if yes, frequency in 24 hour period
Vomiting | 5 days
  yes/no; if yes, frequency in 24 hour period
Elevated gastric residuals | 5 days
  yes/no; if yes, amount (mL) in 24 hour period
Abdominal distention/pain | 5 days
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Krysmaru B AraujoTorres, MD, Study Director — Société des Produits Nestlé (SPN)
Locations (2):
- United States (2):
  - The University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - Le Bonheur Children's Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No